CLINICAL TRIAL: NCT06665035
Title: A Randomized, Age-Descending, Double-Blind, Placebo-Controlled, Phase 3 Trial to Evaluate the Safety and Immunogenicity of 2 Doses of a Subcutaneous Dengue Tetravalent Vaccine (Live, Attenuated) (TDV) Administered Within the Routine Vaccination Schedule of Pediatric Participants ≥6 Months to <21 Months of Age
Brief Title: A Study of 2 Doses of Tetravalent Dengue Vaccine (TDV) in Infants and Toddlers
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: DEN-306; 2023-001084-54 (EudraCT Number)
Record Dates: First submitted 2024-10-29; First posted 2024-10-30 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Dengue Fever
Keywords: Drug Therapy
MeSH Terms: conditions — Dengue

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Cohort 1: Tetravalent Dengue Vaccine (TDV) 0.5 mL (Age group: >=12 to <21 months) (Experimental): Participants with the age group >= 12 to < 21 months receive TDV 0.5 mL subcutaneous (SC) injection, on Day 1 and Day 90.
  Interventions: Biological: TDV
- Cohort 1: Placebo (Age group: >=12 to <21 months) (Experimental): Participants with the age group >= 12 to < 21 months receive placebo (normal saline), SC injection, on Day 1 and Day 90.
  Interventions: Other: Placebo
- Cohort 2: TDV 0.5 mL(Age group: >=6 to <12 months) (Experimental): Participants with the age group >=6 to <12 months receive TDV, 0.5 mL SC injection, on Day 1 and Day 90.
  Interventions: Biological: TDV
- Cohort 2: Placebo (Age group: >=6 to <12 months) (Experimental): Participants with the age group >=6 to <12 months receive placebo (normal saline), SC injection, on Day 1 and Day 90.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: TDV — TDV SC injection.
  Other Names: QDENGA; TAK-003
  Arms: Cohort 1: Tetravalent Dengue Vaccine (TDV) 0.5 mL (Age group: >=12 to <21 months); Cohort 2: TDV 0.5 mL(Age group: >=6 to <12 months)
Other: Placebo — Placebo SC injection.
  Arms: Cohort 1: Placebo (Age group: >=12 to <21 months); Cohort 2: Placebo (Age group: >=6 to <12 months)

SUMMARY:
Dengue fever is caused by an infection with the dengue virus. Vaccination with Dengue Tetravalent Vaccine (TDV) can help prevent dengue fever. The purpose of this study is to collect information of vaccination with TDV when given to children younger than 2 years. The main aims of this study are to learn how safe the vaccine is and how well it works to activate a young child's immune system (this is called immunogenicity). Children between the age of 6 and 21 months will receive two vaccinations with either TDV or placebo 3 months apart. Blood samples will be taken before and after the vaccination as well as throughout the study. These are necessary to check how well the vaccine works to activate the immune system. During the study, participants will visit their study clinic 8 times for vaccinations, blood draws and health checks.

ELIGIBILITY:
Inclusion Criteria

Participant eligibility is determined according to the following criteria:

1. Participant is aged >=6 to <21 months at the time of entry into the trial.
2. Participant is male or female.
3. Participant is in good health at the time of entry into the trial as determined by medical history, physical examination (including vital signs), and the clinical judgment of the investigator.
4. Participant's legally acceptable representative (LAR) has signed and dated a written informed consent form (ICF) and any required privacy authorization prior to the initiation of any trial procedure, and after the nature of the trial has been explained according to local regulatory requirements.
5. The participant and participant's LAR can comply with trial procedures and can be available for the duration of follow-up, according to the LAR.

Exclusion Criteria

Any participant who meets any of the following criteria will not qualify for randomization:

1. Participant has contraindication(s), warning(s) and/or precaution(s) applicable to vaccination with TDV as specified in the investigator's brochure (IB)and/or the approved product label (as applicable) in the participating country.
2. Participant has a known hypersensitivity or allergy to any of the investigational medicinal product (IMP) components (including excipients).
3. Participant has behavioral or cognitive impairment or psychiatric disease that, in the opinion of the investigator, may interfere with the participant's ability to participate in the trial.
4. Participant has a history of progressive or severe neurologic disorder, seizure disorder or neuro-inflammatory disease (example, Guillain-Barré syndrome).
5. Participant has an illness, or history of any illness that, in the opinion of the investigator, might interfere with the results of the trial or pose additional risk to the participant due to involvement in this trial.
6. Participant has a known or suspected impairment/alteration of immune function, including:

   1. Chronic administration of oral and/or parenteral steroids at doses considered sufficiently immunosuppressive (example, >=2 mg/kg [milligrams per kilograms] body weight/day prednisone [or equivalent] for 14 consecutive days, or, >=20 milligram per day [mg/day] prednisone [or equivalent] for >=14 consecutive days) within 60 days prior to Day 1 month 0 (M0) (note: use of corticosteroids by inhaled, intranasal, intraarticular, bursal, tendon injection, or topical routes is allowed).
   2. Receipt of blood, immunoglobulins, blood products, and/or plasma derivatives within the 3 months prior to Day 1 (M0).
   3. Receipt of immunostimulants within 60 days prior to Day 1 (M0).
   4. Immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within 6 months prior to Day 1 (M0).
   5. HIV infection or HIV-related disease.
   6. Hepatitis B virus infection.
   7. Hepatitis C virus infection.
   8. Genetic immunodeficiency.
7. Participant has known or suspected abnormalities of splenic or thymic function.
8. Participant has a known bleeding diathesis, or any condition/medication that may be associated with a prolonged bleeding time.
9. Participant has a serious chronic or progressive disease deemed to be preclusive to trial entry, that is., not medically stable according to the judgment of the investigator.
10. Participant has previously received a vaccination against dengue virus (investigational or licensed).
11. Participant has a clinically significant active infection (as assessed by the investigator) or body temperature greater than (>) 38.0 degrees Celsius (°C) (>100.4 degrees Fahrenheit [°F]) within 3 days of intended IMP administration on Day 1 (M0).
12. Participant has used antipyretics and/or analgesic medications within 24 hours prior to vaccination. The reason for their use (prophylaxis vs treatment) must be documented. Trial entry must be delayed to allow for a full 24 hours to have passed since last use of antipyretics and/or analgesic medications.
13. Participant has received any of the following:

    1. A licensed vaccine within 14 days (for inactivated vaccines) or 28 days (for live vaccines) prior to IMP administration on Day 1 (M0). This includes co-administration with routine vaccines.
    2. A coronavirus vaccine within 14 days prior to IMP administration on Day 1 (M0).
    3. A vaccine authorized for emergency use within 28 days prior to IMP administration on Day 1 (M0).
14. Participant is scheduled to receive any other vaccine within 28 days after IMP administration on Day 1 (M0).
15. Participant is participating in any clinical trial with another investigational product 30 days prior to Day 1 (M0) or plans to participate in another clinical trial at any time during the conduct of this trial.
16. Participant has taken part in any clinical trial of a dengue or other flavivirus (example, West Nile virus) candidate vaccine, except if it is known that the participant received placebo in the trial(s).
17. A first degree relative is involved in the conduct of this trial.

Ages: 6 Months to 20 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 212 (Estimated)
Dates: Start 2025-06-16 (Actual); Primary Completion 2030-03-03 (Estimated); Study Completion 2030-03-03 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Solicited Local (Injection Site) Adverse Events (AEs) Within 7 Days Post Vaccination at Day 1 (Overall and by Severity) | Within 7 Days post-vaccination at Day 1
  Solicited local AEs are injection site pain/tenderness, erythema, and swelling at the vaccination site. All solicited AEs at the injection site will be considered related to the study vaccine administration. The AEs of severity will be graded by investigator as Grade 1: mild, Grade 2: moderate and Grade 3: severe.
Percentage of Participants with Solicited Local (Injection Site) AEs Within 7 Days Post Vaccination at Day 90 (Overall and by Severity) | Within 7 days post-vaccination at Day 90
  Solicited local AEs are injection site pain/tenderness, erythema, and swelling at the vaccination site. All solicited AEs at the injection site will be considered related to the study vaccine administration. The AEs of severity will be graded by investigator as Grade 1: mild, Grade 2: moderate and Grade 3: severe.
Percentage of Participants with Solicited Systemic AEs Within 14 Days Post Vaccination at Day 1 (Overall and by Severity) | Within 14 days post-vaccination at Day 1
  Solicited systemic AEs include fever (body temperature greater than or equal to [>=] 38-degree Celsius [C], drowsiness, irritability/fussiness and loss of appetite. The AEs of severity will be graded by investigator as Grade 1: mild, Grade 2: moderate and Grade 3: severe.
Percentage of Participants with Solicited Systemic AEs Within 14 Days Post Vaccination at Day 90 (Overall and by Severity) | Within 14 days post-vaccination at Day 90
  Solicited systemic AEs include fever (body temperature >= 38 degree (C), drowsiness, irritability/fussiness and loss of appetite. The AEs of severity will be graded by investigator as Grade 1: mild, Grade 2: moderate and Grade 3: severe.
Percentage of Participants with Unsolicited AEs Within 28 Days Post Vaccination at Day 1 | Within 28 days post-vaccination at Day 1
  An unsolicited AE is any AE reported by the participant that is not specified as a solicited AE or is specified as a solicited AE but starts outside the period for reporting a solicited AE (that is, 7 days and 14 days in total including the day IMP administration).
Percentage of Participants with Unsolicited AEs Within 28 Days Post Vaccination at Day 90 | Within 28 days post-vaccination at Day 90
  An unsolicited AE is any AE reported by the participant that is not specified as a solicited AE or is specified as a solicited AE but starts outside the period for reporting a solicited AE (that is, 7 days and 14 days in total including the day of IMP administration).
Percentage of Participants with Medically-attended AEs (MAAEs) | From Day 1 through the end of trial (up to Day 1170)
  MAAEs are defined as AEs leading to an unscheduled visit to or by a healthcare professional including visits to an emergency department (medically attended visits), but not fulfilling seriousness criteria.
Percentage of Participants with Serious Adverse Events (SAEs) | From Day 1 through the end of trial (up to Day 1170)
  SAE is any untoward medical occurrence or effect that at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability / incapacity, is a congenital anomaly / birth defect or is medically important due to other reasons than the above-mentioned criteria.
Geometric Mean Titers (GMTs) of Neutralizing Antibodies by Microneutralization Test (MNT) for Each of 4 Dengue Virus Serotypes at Day 120 | Day 120
  GMTs of neutralizing antibodies will be measured by MNT against 4 dengue virus serotypes. The 4 dengue virus serotypes are dengue virus (DENV-1, DENV-2, DENV-3 and DENV-4) will be reported.

SECONDARY OUTCOMES:
GMTs of Neutralizing Antibodies by MNT for Each of the 4 Dengue Virus Serotypes | Day 1, Day 30, Day 270, Day 450, Day 810 and Day 1170
  GMTs of neutralizing antibodies will be measured by MNT against 4 dengue virus serotypes. The 4 dengue virus serotypes are DENV-1, DENV-2, DENV-3 and DENV-4.
Seropositivity Rates for 4 Dengue Virus Serotypes | Day 1, Day 30, Day 120, Day 270, Day 450, Day 810 and Day 1170
  Seropositive rate is defined the percentage of participants with MNT titer >=10 against each of the four dengue virus serotypes. The four dengue virus serotypes (DENV-1, DENV-2, DENV-3 and DENV-4) will be reported.
Seropositivity Rates For Multiple (2, 3, or 4) Dengue Virus Serotypes | Day 1, Day 30, Day 120, Day 270, Day 450, Day 810 and Day 1170
  Seropositive rate is defined the percentage of participants with MNT titer >=10 against multiple (2, 3, or 4) dengue virus serotypes. The 4 dengue virus serotypes are DENV-1, DENV-2, DENV-3 and DENV-4.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director Study Director, Study Director — Takeda
Locations (4):
- Colombia (2):
  - Clinica de la Costa Ltda, Barranquilla, Atlántico
  - Centro de Estudios en Infectologia Pediatrica S.A.S, Cali, Valle del Cauca Department
- Thailand (2):
  - King Chulalongkorn Memorial Hospital, Pathum Wan, Bangkok
  - Thammasat University Hospital, Khlong Luang, Changwat Pathum Thani

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/